CLINICAL TRIAL: NCT01139697
Title: Hair Cortisol and Testosterone Levels and Their Correlation With Heart Failure Status in Patients With Chronic Congestive Heart Failure
Brief Title: Hair Cortisol and Testosterone in Heart Failure
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: cortest-chf-1
Record Dates: First submitted 2010-05-20; First posted 2010-06-08 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Systolic Heart Failure
Keywords: Heart failure; Cortisol; Testosterone
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hair samples for the measurment of cortisol and testosterone
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with systolic heart failure: Patients with systolic heart failure defined as ejection fraction <45%
  Interventions: Other: Hair sampling

INTERVENTIONS:
Other: Hair sampling — Hair sampling for the measurement of cortisol and testosterone

SUMMARY:
The purpose of this study is to determine whether hair cortisol and testosterone levels correlate with heart failure status in patient with chronic congestive heart failure.

DETAILED DESCRIPTION:
Progression of chronic congestive heart failure (CHF) is associated with abnormal secretion of several hormones including glucocorticoids and testosterone.

A single study of patients with chronic heart failure has demonstrated that higher serum levels of cortisol are independent predictors of increased mortality risk. However, this study included patients with heart failure who were admitted to the hospital due to other causes and it might be speculated that the single serum cortisol measurement taken may have been influenced by the acute illness or by the emotional stress associated with the admission itself.

Currently, there are several modalities for measuring cortisol levels including serum, urinary and salivary techniques. However, all these methods represent indicators of acute cortisol secretion and do not reflect accumulation of the hormone over time. Recently there has been a growing interest in measuring hair cortisol level. Hair grows approximately 1 centimeter per month and therefore hair analysis accurately reflects long-term endogenous production of cortisol. This provides for the first time a reliable mode for the measurement of the accumulation of cortisol over time. We have recently demonstrated higher hair cortisol levels in patients with acute myocardial infarction compared with controls (the manuscript has been submitted for publication). Regarding testosterone, several studies have recently demonstrated lower free serum testosterone levels in patients with heart failure compared with controls. Furthermore, Serum testosterone levels were inversely correlated with heart failure status.

The longitudinal assessment of cortisol and testosterone levels over time using the hair technique may be superior to a single random serum sample for the assessment of chronic heart failure status and prognosis.

If indeed, hair cortisol and testosterone levels would correlate with heart failure status, they may be used as a quantitative mode for clinical follow-up of CHF patients (similar to the role of HbA1C in the follow-up of diabetic patients). However this hypothesis has not yet been evaluated

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age >18
* Left ventricular (LV) systolic function (EF<45 per echocardiography)

Exclusion Criteria:

* Any corticosteroid treatment in the last 6 months
* Any treatment with testosterone in the last 6 months
* Diagnosis or Cushing's or Addison's disease
* Any hospital admission within 3 months prior to enrollment
* Inability to sign inform consent
* Patients with moderate or severe aortic stenosis
* Inability to provide 3 cm hair sample from vertex posterior.
* Dyed hair
* Morbid obesity (BMI>35)
* Any symptomatic chronic lung disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systolic heart failure from the out-patient clinic at the Meir Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-08

PRIMARY OUTCOMES:
Correlation of hair cortisol and testosterone with heart failure status | One year
  Ccorrelation of hair cortisol and testosterone with clinical and laboratory parameters that their correlation with heart failure status is well established including:
  1. Ejection fraction as assessed by echo-doppler.
  2. Physical capacity as assessed by stress test.
  3. Serum levels of hs-CRP, NT-proBNP. 4)1 year mortality
  5)hospital admissions after 6 and 12 months

SECONDARY OUTCOMES:
Mortality | 6 and 12 months
  The association of hair cortisol and testosterone with mortality
Hospital adMissions | 6 and 12 months
  The correlation of hair cortisol and testosterone with hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: David Pereg, MD, Principal Investigator — Cardiology department, Meir Medical Center; Morris Mosseri, MD, Principal Investigator — Cardiology departement, Meir medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Background] Guder G, Bauersachs J, Frantz S, Weismann D, Allolio B, Ertl G, Angermann CE, Stork S. Complementary and incremental mortality risk prediction by cortisol and aldosterone in chronic heart failure. Circulation. 2007 Apr 3;115(13):1754-61. doi: 10.1161/CIRCULATIONAHA.106.653964. Epub 2007 Mar 19. PMID 17372171
- [Background] Sauve B, Koren G, Walsh G, Tokmakejian S, Van Uum SH. Measurement of cortisol in human hair as a biomarker of systemic exposure. Clin Invest Med. 2007;30(5):E183-91. doi: 10.25011/cim.v30i5.2894. PMID 17892760
- [Background] Van Uum SH, Sauve B, Fraser LA, Morley-Forster P, Paul TL, Koren G. Elevated content of cortisol in hair of patients with severe chronic pain: a novel biomarker for stress. Stress. 2008 Nov;11(6):483-8. doi: 10.1080/10253890801887388. PMID 18609301
- [Background] Brotman DJ, Golden SH, Wittstein IS. The cardiovascular toll of stress. Lancet. 2007 Sep 22;370(9592):1089-100. doi: 10.1016/S0140-6736(07)61305-1. PMID 17822755
- [Background] Guder G, Frantz S, Bauersachs J, Allolio B, Ertl G, Angermann CE, Stork S. Low circulating androgens and mortality risk in heart failure. Heart. 2010 Apr;96(7):504-9. doi: 10.1136/hrt.2009.181065. Epub 2009 Oct 28. PMID 19875366
- [Background] Jankowska EA, Filippatos G, Ponikowska B, Borodulin-Nadzieja L, Anker SD, Banasiak W, Poole-Wilson PA, Ponikowski P. Reduction in circulating testosterone relates to exercise capacity in men with chronic heart failure. J Card Fail. 2009 Jun;15(5):442-50. doi: 10.1016/j.cardfail.2008.12.011. Epub 2009 Feb 10. PMID 19477405